CLINICAL TRIAL: NCT06657651
Title: Autogenous Dentine Derived Barrier Membrane Versus Extended Platelet Rich Fibrin Membrane in Immediate Implant Placement
Brief Title: IMMEDIATE IMPLANT With Different Types of Membranes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A06030240S
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Tooth Extraction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant with dentin-derived membrane (Experimental)
  Interventions: Procedure: immediate implant placement with dentin-derived membrane
- immediate implant with extended platelet rich fibrin membrane (Experimental)
  Interventions: Procedure: immediate implant with extended platelet rich fibrin membrane

INTERVENTIONS:
Procedure: immediate implant placement with dentin-derived membrane — immediate implant placement with dentin-derived membrane and allograft in mandibular molar area
  Arms: immediate implant with dentin-derived membrane
Procedure: immediate implant with extended platelet rich fibrin membrane — immediate implant with extended platelet rich fibrin membrane and allograft in mandibular molar area
  Arms: immediate implant with extended platelet rich fibrin membrane

SUMMARY:
forty patients will be selected from the outpatient's clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University for replacement of non-restorable tooth in posterior mandibular area.

Patients' Grouping:

The patients will be randomly divided into two equal uniform groups each consists of 20 patients:

Group A:

20 patients with non-restorable mandibular molar tooth will be treated with an immediately placed dental implant in conjunction with a dentin-derived membrane from the extracted tooth.

Group B:

20 patients with non-restorable mandibular molar tooth will be treated with an immediately placed dental implant in conjunction with extended platelet rich fibrin membrane.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Non-restorable mandibular molar tooth that needs dental extraction & guided bone regeneration for immediate implant placement.
* Acceptable inter-arch space for the future prosthesis.
* Patient medically free from systemic diseases that absolutely contraindicate implant surgery.
* Cooperative patient with high motivation and acceptable oral hygiene.
* Free from history of bruxism / parafunctional habits.

Exclusion Criteria:

* Local and / or systemic conditions that interfere with the procedure.
* Smokers.
* Pregnancy.
* Uncooperative patients.
* Patient had undergone in the past 12 months radiation therapy to the head and neck area.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Implant stability | 1 year
  Osstell will be used to record implant stability at the placement time, 3, 6 and 12 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Elsheikh, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No